CLINICAL TRIAL: NCT06881836
Title: A Phase II, 26-week, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of ONO-2020 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Study of ONO-2020 in Participants With Mild to Moderate Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONO-2020-02; jRCT2031240712 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-03-02; First posted 2025-03-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; mild to moderate Alzheimer Disease; Dementia; ONO-2020
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ONO-2020 Dose 1 (Experimental): Participants will receive ONO-2020 Dose 1 administered orally, once a day (QD) for 26 weeks.
  Interventions: Drug: ONO-2020
- ONO-2020 Dose 2 (Experimental): Participants will receive ONO-2020 Dose 2 administered orally, once a day (QD) for 26 weeks.
  Interventions: Drug: ONO-2020
- Placebo (Placebo Comparator): Participants will receive Placebo administered orally, once a day (QD) for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-2020 — ONO-2020 group: Two ONO-2020 tablets will be orally administered once daily.
  Arms: ONO-2020 Dose 1; ONO-2020 Dose 2
Drug: Placebo — Placebo group: Two ONO-2020 placebo tablets will be orally administered once daily.
  Arms: Placebo

SUMMARY:
This is a Phase 2, double-blind, parallel-group, placebo-controlled study to assess safety, tolerability, pharmacokinetics, and efficacy of ONO-2020 in participants with mild to moderate Alzheimer's disease (AD). This study aims to determine whether administering ONO-2020, an epigenetic regulator, may improve cognitive functions like memory and cognition in individuals with Alzheimer's disease dementia.

DETAILED DESCRIPTION:
In the study, participants will undergo a screening period of up to 6 weeks (42 days). Eligible participants will be assigned to receive one of 2 dose levels of ONO-2020 or placebo control arm. ONO-2020 or placebo will be administered orally QD for 26 weeks. All participants who received study intervention will be followed up for 4 weeks after treatment discontinuation. The target sample size is 240 participants , out of which up to 45 participants will undergo additional special CSF biomarker evaluation. After enrollment, participants will be randomized in a 1:1:1 ratio to one of 3 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of Alzheimer's disease according to the recommendations from the revised criteria for diagnosis and staging of Alzheimer's disease: Alzheimer's Association Workgroup , along with any positive AD-specific biomarker results (abnormal Core 1 or Core 2 biomarkers) from a previous diagnosis or at screening.
2. Have a previous MRI or CT scan of the brain, which was performed within 1 year prior to enrollment in the study, to confirm that more recent neurological events (e.g., stroke) would not potentially constitute a confounder in the assessment of the etiology of the participant's cognitive status.
3. MMSE score of 15 to 24, inclusive, and MMSE score cannot deviate more than 3 points in either direction between the screening and baseline visits.
4. AD numeric clinical stage 4 or stage 5 based on NIA-AA criteria 2024, at screening and baseline visits
5. Participants receiving concurrent AD treatment (acetylcholinesterase inhibitors and /or memantine) must be on a stable dose for at least 90 days prior to randomization, and the participant must be willing to remain on the same dose for the duration of the study.
6. Have the ability to comply with procedures for cognitive and other tests in the opinion of the investigator
7. If female, postmenopausal for at least 1 year
8. Non-vasectomized male participants with female partners of childbearing potential must agree to use an effective method of contraception from dosing on Day 1 until 3 months after the last administration of study intervention and agree not to donate sperm until 3 months after the last administration of study intervention.
9. Participant must have a Caregiver who has frequent contact with the participant (defined as at least 8 hours per week spread across 3~4 visits per week) to provide support to the participant to ensure compliance with study requirements. The Caregiver must be willing to consent to participate in this study, to provide a rating of the extent and severity of change of the participant's memory, problem-solving abilities, or activities of daily living from prior abilities.
10. General health status acceptable for participation in the study, and the participant must be able to ingest pills.
11. Participant and his/her Caregiver have provided full written informed consent prior to the performance of any protocol-specified procedure; or if a participant is unable to provide informed consent due to cognitive status, he/she has provided assent, and a legally acceptable representative (LAR) has provided full written informed consent on behalf of the participant.

Exclusion Criteria:

1. Participants with dementia or other memory impairment not due to Alzheimer's disease, including, but not limited to, dementia with Lewy bodies, vascular dementia, Parkinson's disease, Huntington disease, corticobasal degeneration, Creutzfeldt-Jakob disease, progressive supranuclear palsy, frontotemporal degeneration, normal pressure hydrocephalus, hypoxia, severe sleep apnea or other chronic sleep disturbance, or baseline intellectual disability.
2. Participants with a history of stroke, well-documented transient ischemic attack, or pulmonary or cerebral embolism.
3. History of significant psychiatric illness such as schizophrenia or bipolar affective disorder, or history or current major depressive disorder in the past year and any other significant psychiatric illness that in the opinion of the investigator could interfere with participation in the study.
4. Participants with delirium or history of delirium within the 30 days prior to the screening visit.
5. Have suicide ideation according to the investigator's clinical judgment as per the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening or have made a suicide attempt in the 6 months prior to screening.
6. Clinically significant ECG abnormality as judged by the investigator.
7. Confirmed absolute QTcF >450 msec for males or >470 msec for females.
8. Positive results at screening for active viral infections that include human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) RNA PCR test.
9. Participants with total bilirubin, alanine transaminase (ALT) or aspartate transaminase (AST) greater than 1.5×upper limit of normal (ULN), or international normalized ratio (INR) greater than 1.7 at screening.
10. Participants with estimated creatinine clearance (CrCL, Cockcroft-Gault equation) ≤30 mL/min at screening.
11. Participants with a history of treatment, and/or current treatment, with anti-Aβ antibodies
12. Changes in any medications that, in the opinion of the investigator, may potentially impair participants' ability to perform cognitive testing or study procedures during the study period (from Screening to EOT), and their dosing should be stable for at least 1 month before Screening (such as benzodiazepines and sedatives/hypnotics). All concomitant medications must be kept as stable as medically possible during the study.
13. Participants who have taken any investigational products, or used investigational medical devices, within 3 months or five half-lives of the therapy (whichever is longer) with respect to first dosing and throughout the study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment emergent adverse events (TEAEs) | From baseline up to 26 weeks
  The number and percentage of subjects reporting each TEAE will be summarized by both system organ class (SOC) and preferred term (PT).
Clinically abnormal findings in Columbia Suicide Severity Rating Scale (C-SSRS) | From baseline up to 26 weeks
  The number and percentage of subjects with clinically abnormal finding will be tabulated at each time point.
Change from baseline through week 26 in Alzheimer's Disease Assessment Scale-Cognitive Subscale 12 (ADAS-cog 12) score | From baseline up to 26 weeks

SECONDARY OUTCOMES:
Change from baseline through week 26 in ADAS-cog 12 score in mild AD participants | From baseline up to 26 weeks
Change from baseline through week 26 in ADAS-cog 12 score in moderate AD participants | From baseline up to 26 weeks
Change from baseline through week 26 in ADAS-cog 11 and 13 scores | From baseline up to 26 weeks
Change from baseline through week 26 in Alzheimer's Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL) score | From baseline up to 26 weeks
Change from baseline through week 26 in Quick Dementia Rating System (QDRS) | From baseline up to 26 weeks
Change from baseline through week 26 in Mini-Mental State Examination (MMSE) score | From baseline up to 26 weeks
Change from baseline through week 26 in Neuropsychiatric Inventory Questionnaire (NPI-Q) | From baseline up to 26 weeks
Change from baseline through week 26 in Quality of Life-Alzheimer's Disease (QoL-AD) Scale | From baseline up to 26 weeks
Change from baseline through week 26 in Zarit Burden Interview Scale (ZBI) | From baseline up to 26 weeks
Change in plasma concentration of ONO-2020 by dose level and time point | Day 1, Week 2, Week 10, and Week 26
  The plasma concentrations of ONO-2020 will be listed, and descriptive summary statistics of them will be calculated by dose level and time point.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (96):
- United States (76):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute (BAI), Phoenix, Arizona
  - Clinical Endpoints, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Center for Neurosciences-Research, Tucson, Arizona
  - Profound Research LLC at The Neurology Center of Southern California, Carlsbad, California
  - Neurology Center of North Orange County, Fullerton, California
  - Stanford University, Palo Alto, California
  - Sunwise Clinical Research, Walnut Creek, California
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Brain Matters Research, Delray Beach, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Premier Clinical Research Institute; Inc., Miami, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Orlando, Orlando, Florida
  - Accel Research Sites - Brain and Spine Institute, Port Orange, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Charter Research - The Villages, The Villages, Florida
  - Conquest Research LLC, Winter Park, Florida
  - Sandhill Research, LLC d/b/a Accel Research Sites - NeuroStudies CRU, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Re:Cognition Health-Chicago, Chicago, Illinois
  - Charter Research - Chicago, Chicago, Illinois
  - Ascension Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - University of Kansas Medical Center, Fairway, Kansas
  - Univ of Kentucky Sanders-Brown Center on Aging, Lexington, Kentucky
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Research, Methuen, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ (CenExel AMRI), Toms River, New Jersey
  - Advanced Clinical Institute Inc., West Long Branch, New Jersey
  - Integrative Clinical Trials, Brooklyn, New York
  - University at Buffalo, Buffalo, New York
  - Velocity Clinical Research; Syracuse, East Syracuse, New York
  - The Feinstein Institutes for Medical Research, Manhasset, New York
  - NYU Center for Cognitive Neurology, New York, New York
  - AD-CARE; University of Rochester, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Eximia Research-Raleigh, Raleigh, North Carolina
  - Velocity Clinical Research at Raleigh Neurology, Raleigh, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Neurology Diagnostics Research, Dayton, Ohio
  - Neuro Behavioral Clinical Research, Inc., North Canton, Ohio
  - Neural Net Research / Center for Cognitive Health, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Penn Medicine, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Alliance for Multispecialty Research;LLC-Knoxville, Knoxville, Tennessee
  - Vanderbilt UMC-Cognitive Med, Nashville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Horizon Clinical Research Group, Cypress, Texas
  - Texas Neurology, Dallas, Texas
  - FutureSearch Trials of Dallas LLC, Dallas, Texas
  - Re:Cognition Health - Fort Worth, Fort Worth, Texas
  - Re:Cognition Health - Houston, Houston, Texas
  - Olympus Clinical Research - Katy, Katy, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Wasatch Clinical Research; LLC, Salt Lake City, Utah
  - Re:Cognition Health - Fairfax, Fairfax, Virginia
  - Sentara Neurology Specialists, Norfolk, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Kingfisher Cooperative; LLC, Spokane, Washington
- Japan (20):
  - National Center for Geriatrics and Gerontology, Aichi
  - Inage Neurology and Memory Clinic, Chiba
  - Mabashi Clinic, Chiba
  - Southern Tohoku Medical Clinic, Fukushima
  - Ikuseikai Shinozuka Hospital, Gunma
  - Imon Yukari Neurology Clinic, Hiroshima
  - NHO Hiroshima-Nishi Medical Center, Hiroshima
  - Himeji Central Hospital Clinic, Hyōgo
  - Kobe City Medical Center General Hospital, Hyōgo
  - Memory Clinic Toride, Ibaraki
  - Kagawa Prefectural Central Hospital, Kagawa
  - Meiwakai Izaki Clinic, Nagasaki
  - Katayama Medical Clinic, Okayama
  - Takesato Hospital, Saitama
  - Jichiidai Station Brain Clinic, Tochigi
  - Ichiekai Itsuki Hospital, Tokushima
  - Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital, Tokyo
  - Memory Clinic Ochanomizu, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Metropolitan Institute for Geriatrics and Gerontology, Tokyo

IPD SHARING:
Plan to Share IPD: No